CLINICAL TRIAL: NCT06638632
Title: Helping Patients, Families, and Clinicians Make Shared Decisions About Therapies for Dementia
Brief Title: Decision Aid for Dementia Therapies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-0866; NIA Grant#: R21AG088955 (Other Grant/Funding Number: NIA)
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Decision Aids
Keywords: Lecanemab
MeSH Terms: conditions — Dementia | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: This is an iterative, user-centered design process. Therefore, patients and care partners will receive iterations of the decision aid as updates are made to it.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Aid (Experimental): Participants provide feedback on the development of a decision aid for dementia therapies.
  Interventions: Behavioral: Decision aid

INTERVENTIONS:
Behavioral: Decision aid — Patients with dementia and care partners will receive an iteration of the decision aid and provide feedback.

SUMMARY:
The purpose of this study is to develop a decision aid to support patients and families making decisions about medications for dementia.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* UCHealth patient
* Ages 18 y/o and above
* Documented neurocognitive deficits suggestive of mild cognitive impairment or early dementia as determined by their treating clinician.
* English or Spanish speaking

Caregiver:

* Ages 18 y/o and above
* Identified by the study participant as the person who helps the most with their medical care outside the hospital or clinic.
* English or Spanish speaking

Clinicians:

* Neurologists, primary care clinicians, pharmacists, or psychologists involved in dementia decision-making.
* English or Spanish speaking

Exclusion Criteria:

Patients:

* Not English or Spanish-speaking
* Neurocognitive deficits suggestive of moderate or severe cognitive impairment or late stage dementia.
* Not able to consent for themselves

Caregiver:

* Ages 17 y/o and below
* Not English or Spanish-speaking

Clinicians:

* Neurologists, primary care clinicians, pharmacists, or psychologists involved in dementia decision-making.
* English or Spanish-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict | From enrollment at start of year 2 to the end of year 2
  To access the preliminary efficacy on decisional conflict including personal perceptions of uncertainty in choosing options, factors that contribute to feelings of uncertainty and effective decision making.
  Decisional Conflict Scale - Higher numbers mean more uncertainty. O'Connor, A. M. (1995). Validation of a decisional conflict scale. Medical decision making, 15(1), 25-30. https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decisional_Conflict.pdf
Shared Decision Making | From enrollment at start of year 2 to the end of year 2
  To determine the extent that health care providers engage with patients as a part of their shared decision making, specifically looking at the discussion of treatment options and their pros and cons as well as the patient's preferences.
  Shared Decision Making Process Scale - Higher numbers mean more shared decision making. https://mghdecisionsciences.org/tools-training/sdm-process-survey/
Decisional Self-Efficacy | From enrollment at start of year 2 to the end of year 2
  To determine the patient's perception of their self-efficacy in decision making including measuring their self-confidence in their ability to make decisions.
  Decision Self-Efficacy Scale where higher numbers mean they patient has a higher perception of self-efficacy.
  https://decisionaid.ohri.ca/docs/develop/Tools/Decision_SelfEfficacy.pdf

CONTACTS AND LOCATIONS:
Overall Officials: Dan Matlock, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elwyn G, Frosch D, Volandes AE, Edwards A, Montori VM. Investing in deliberation: a definition and classification of decision support interventions for people facing difficult health decisions. Med Decis Making. 2010 Nov-Dec;30(6):701-11. doi: 10.1177/0272989X10386231. Epub 2010 Nov 18. PMID 21088131
- [Background] van Dyck CH, Swanson CJ, Aisen P, Bateman RJ, Chen C, Gee M, Kanekiyo M, Li D, Reyderman L, Cohen S, Froelich L, Katayama S, Sabbagh M, Vellas B, Watson D, Dhadda S, Irizarry M, Kramer LD, Iwatsubo T. Lecanemab in Early Alzheimer's Disease. N Engl J Med. 2023 Jan 5;388(1):9-21. doi: 10.1056/NEJMoa2212948. Epub 2022 Nov 29. PMID 36449413